CLINICAL TRIAL: NCT02465385
Title: Single-dose Linaclotide for Capsule Endoscopy Preparation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, R. Ann Hays, MD, Assistant Professor, Gastroenterology, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 17803
Record Dates: First submitted 2015-05-27; First posted 2015-06-08 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Crohn's; Ulcerative Colitis; Gastrointestinal Bleeding
MeSH Terms: conditions — Colitis, Ulcerative; Gastrointestinal Hemorrhage | interventions — linaclotide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Linaclotide 290mcg
  Interventions: Drug: Linaclotide

INTERVENTIONS:
Drug: Linaclotide — Every participant with be given 290 mcg of linaclotide 1 hour prior to receiving their capsule, in place of the standard (golytely) preparation
  Other Names: Linzess

SUMMARY:
Video capsule endoscopy is an important procedure that can be used by doctors to find abnormalities in the small intestine, especially those that can cause bleeding. The procedure uses a tiny wireless camera to take pictures of the digestive tract. The camera sits inside a vitamin-sized capsule that a person can swallow. As the capsule travels through the digestive tract, the camera takes thousands of pictures that are transmitted to a recorder worn on a belt around a person's waist or over his/her shoulder. However, abnormalities can be missed partly because the normal dark liquids present in the intestine can prevent abnormalities from being recorded, hiding them from the physician who reviews the video.

The current method used to clear these dark liquids from your small intestine is to follow a clear liquid diet and drink approximately 2 quarts of polyethylene glycol (Golytely®) the day before the video endoscopy and take simethicone (a medication used to treat symptoms of gas such as uncomfortable or painful pressure, fullness, and bloating) the morning of the test.

Some of the current preparations to clear these dark liquids are not able to entirely prevent abnormalities from being missed and most have an unpleasant taste or involve drinking a lot of fluid.

Linaclotide (Linzess®) is a medication approved by the Food and Drug Administration (FDA) for the treatment of constipation and irritable bowel syndrome. It is not approved by the FDA for use as an aid for clearing dark liquid from the small intestine prior to a video endoscopy.

A recent presentation at a medical meeting proposed using one-dose of linaclotide (Linzess®) to improve cleansing of the small intestine for capsule endoscopy preparation to supplement fasting and clear liquid diet.

This report claimed a noticeably better quality of small intestine cleansing and a 20% shorter transit time for the capsule by taking one dose of linaclotide one hour before patients swallowed the video capsule.

The purpose of this study is to assess the use of one dose of linaclotide in terms of the total time it takes the capsule to move through the small bowel, and image quality as compared to the current method. The results of this study will be compared to previous patients who drank the preparation that is currently used

DETAILED DESCRIPTION:
Video capsule endoscopy is an important modality for detection of lesions in the small intestine. It is particularly helpful in patients with occult sources of gastrointestinal bleeding, suspected Crohn's disease, ulcerative jejunitis, and in cases where a small intestinal neoplasm is suspected. Despite advances in technique and equipment, significant limitations remain in obtaining adequate visualization due to dark bilious fluid that obscures the mucosa. Furthermore, limitations of battery technology mean that in approximately 16.5% of studies the capsule will fail to visualize the entire small bowel. Numerous methods of bowel preparation have been used for capsule endoscopy. To date, all of them are unpleasant/have significant side effects. This is particularly onerous given that the majority has already had a similar but more extensive preparation for colonoscopy. Furthermore, overall efficacy is varied, and the preparation frequently remains suboptimal. The University of Virginia Health System Motility Lab uses a current regimen of 2000 mL of golytely and simethicone, but incomplete and partially occluded portions of the small bowel remain persistent clinical issues. Nearly one in five studies may ultimately have to be repeated as a result.

A recent presentation by Ira J. Schmelkin, M.D. proposed the use of single-dose linaclotide for capsule endoscopy preparation to supplement fasting and clear liquid diet. In an uncontrolled series, he noted a clinically significant improvement in preparation quality and a 20% shorter transit time (compared with published norms) with one higher range dose of linaclotide an hour prior to endoscopy. Linaclotide is guanylate cyclase-C that acts on the luminal surface of the intestinal epithelium thereby stimulating secretion of chloride and bicarbonate into the intestinal lumen, resulting in increased intestinal fluid and increased motility. The increased motility and secretion throughout the gastrointestinal tract make it a potentially useful agent to decrease capsule transit time and decrease the amount of dark small intestine fluid, thereby improving capsule endoscopy yield. Initial reports suggest that linoclotide is generally well tolerated, with the primary side effect of diarrhea. The investigators propose to study the use of a single dose for capsule endoscopy preparation.

The hypothesis is that single-dose linaclotide will lead to significantly decreased transit time and improved small bowel visualization quality when compared to controls using polyethylene glycol and simethicone (standard of care).

The investigators propose to prospectively enroll approximately 30 patients as subjects, who will receive a single dose of 290mcg one hour prior to capsule endoscopy. This was calculated using power calculations from values of the Viazis study, who noted an average transit time of approximately 290 minutes, compared with approximately 190 minutes in the data from Schmelkin. Given the standard deviation of approximately 90 minutes in Viazis, power calculation with an alpha of 0.05 and a beta of 0.80 would require 18 subjects per group. The investigators will target 30 to allow for dropouts and to allow the use of statistics pertaining to large (approximately 30 and up) numbers of subjects.

All adult patients undergoing capsule endoscopy (with the exception of certain criteria, such as severe gastroparesis, pregnancy, non-English speaking, prisoners, those unable to give consent, prior small intestinal resection) will be approached sequentially until completion of the study. These will be matched 1:1 with historic controls selected at random from cases in the prior three years. The same exclusion criteria will be applied to both groups. There will be two primary outcomes: total transit time and rated overall mucosal visualization (categorized as ideal, good, inadequate or poor/needs repetition). Primary analysis will presume no confounding and use a t-test and chi-square, respectively. Should the groups prove significantly different, the investigators also plan to use adjusted analysis. The investigators will plan to collect BMI, history of reflux, age, sex, gastroparesis, diabetes, narcotic use, other conditions e.g. Parkinson's, lupus, scleroderma as these may affect transit time for the historic controls.

Two gastrointestinal fellows or attending level gastroenterologists will perform the scoring of the images recorded during the capsule endoscopy in a blinded manner. Secondarily, the investigators will also look at the percentage of capsule endoscopies detecting a culprit lesion, and the percentage of failed (incomplete) studies.

ELIGIBILITY:
Inclusion Criteria:

* Schedule for video endoscopy at UVHS
* Ability to speak, read and write English
* Age >18
* Able to provide consent

Exclusion Criteria:

* Prisoner
* Woman who is currently pregnant or breastfeeding
* Allergy to linaclotide
* Patients with known or suspected mechanical gastrointestinal obstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Small bowel transit time | 10 hours post-dose
  The time of transit will be reviewed on the following day after the study. The data is collected when the capsule is finished recording, approximately 10 hours post-dose

SECONDARY OUTCOMES:
Overall mucosal visualization on the recorded images as rated by an expert reviewer and graded on a 5-point likert scale. | 10 hours post-dose
  The mucosal visualization will be reviewed on the following day after the study. The data is collected when the capsule is finished recording, approximately 10 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Hays, MD, Principal Investigator — Assistant professor
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Derived] Stein DJ, Copland A, McDaniel D, Hays RA. Single-Dose Linaclotide Is Equal in Efficacy to Polyethylene Glycol for Bowel Preparation Prior to Capsule Endoscopy. Dig Dis. 2019;37(4):297-302. doi: 10.1159/000496350. Epub 2019 Feb 7. PMID 30731474